CLINICAL TRIAL: NCT01373801
Title: THE EFFICACY AND SAFETY OF HEMCON© BANDAGE FOLLOWING SURGICAL REPAIR IN MANAGEMENT OF POSTPARTUM BLEEDING DUE TO THE MULTIPLE VAGINAL LACERATIONS
Brief Title: Hemcon© Bandage for Postpartum Bleeding Due to the Multiple Vaginal Lacerations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Collaborators: HemCon Medical Technologies, Inc (Industry)
Responsible Party: Prof. Arnon Wiznitzer, Head of Obstetrics and Gynecology Division, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sor517911ctil
Record Dates: First submitted 2011-06-13; First posted 2011-06-15 (Estimated); Last update posted 2011-08-10 (Estimated); Status verified 2011-04

CONDITIONS: Postpartum Bleeding; Vaginal Lacerations; Cervical Lacerations
Keywords: Postpartum women, after surgical repair of vaginal and cervical lacerations
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator)
  Interventions: Device: The HemCon GuardaCare; Device: Control
- GuardaCare (Experimental)
  Interventions: Device: The HemCon GuardaCare

INTERVENTIONS:
Device: The HemCon GuardaCare — The HemCon GuardaCare (HemCon Medical Technologies Inc., Portland, OR) is a hemostatic dressing made of chitosan, a complex carbohydrate derived from chitin from shellfish and is designed as a hemostatic dressing, and a topical antimicrobial dressing. GuardaCare contains no pro-clotting agents, providing a safe and localized hemostatic solution and is latex free and sterile.
Device: Control — Standard packing gauze roll bandage.
  Arms: Control

SUMMARY:
The objective of the study is to assess the safety and efficacy of the HemCon GuardaCareXR compared to standard bandaging in subjects with post partum hemorrhage as a result of cervical and vaginal lacerations. The primary endpoint will be a cessation of bleeding at 30 minutes after insertion of the dressing.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Age≥18 year
3. Two or more 2nd degree vaginal lacerations , 3rd degree vaginal lacerations and cervical laceration

Exclusion Criteria:

1. Subjects undertaking anticoagulation treatment
2. Pre-existing coagulopathy
3. Massive uncontrolled bleeding requiring blood transfusions/urgent vascular surgery.
4. Systolic blood pressure <90mmHg
5. Shellfish allergy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Cessation of bleeding after a 30 minutes | 30 minutes
  The primary endpoint is a cessation of bleeding after a 30 minute period. Evaluation of bleeding will be performed by an independent evaluator, who will determine if the bleeding has stopped.

SECONDARY OUTCOMES:
Safety composite endpoint | 7 days
  Rate of the safety composite (any of the following):
  1. Anaphylaxis or allergic reaction
  2. Recurrent Hospitalization
  3. Serious adverse events
  4. Need for the repeated surgical intervention
  5. Need for blood products transfusion
  6. Local Infection In addition individual rates of the components will be reported
Device Success | 6 hours
  Device success defined as a cessation of bleeding at 6 hours using only the allocated device.
Procedural success | 6 hours
  Procedural success defined as a cessation of bleeding at 6 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Wiznitzer, M.D, Principal Investigator — Soroka University Medical Center; Victor Novack, M.D. PhD, Principal Investigator — Soroka University Medical Center
Locations (1):
- OB\GYN Soroka University Medical Center, Beersheba, Israel